CLINICAL TRIAL: NCT00780429
Title: Evaluation of Pharmacokinetic and Pharmacodynamic Parameters in Renal Transplant Patients Receiving Mycophenolic Acid and Stable for at Least 3 Months
Brief Title: Pharmacokinetics and Pharmacodynamics of MPA in Stable Renal Transplant Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Prof. Antonio Dal Canton, IRCCS Fondazione Policlinico San Matteo
Other Study IDs: 06/2006/REVO
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Kidney Transplantation
Keywords: kidney; transplant; Mycophenolic acid; Inosine monophosphate dehydrogenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: MMF+cyclosporine
- 2: MMF+tacrolimus
- 3: MMF+sirolimus

SUMMARY:
Study of the pharmacokinetic and pharmacodynamic variability of mycophenolate mofetil in renal transplant patients already on long-term MMF treatment (at least 6 months post-transplant; at least 3 months in therapy).

Study hypothesis: to investigate whether long-term MMF therapy alters IMPDH biological activity and if there are any correlations with the risk of AR.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients
* Age range: 18-70
* Patients taking MMF
* Able to understand and sign an informed consent

Exclusion Criteria:

* Active myelodepression
* Systemic infections or other that may affect MMF absorption
* Pregnancy/breastfeeding
* (History of) cancer
* Drug abuse, psychiatric conditions
* Already enrolled in other clinical trials or participation ended less than one month earlier
* Known sensitivity to polysorbate 80 or MMF

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female renal transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Policlinico San Matteo, Pavia, Italy